CLINICAL TRIAL: NCT07175688
Title: Study of Metabolic Associated Fatty Liver Disease (MAFLD) and Pancreatic Steatosis in Obese Versus Lean Chronic Hepatitis B Patients
Brief Title: Metabolic Associated Fatty Liver Disease and Pancreatic Steatosis in Obese Versus Lean Chronic Hepatitis B Patients
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Samar Hosny Salama, Assistant lecturer of Tropical Medicine and Infectious Diseases, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 35454/4/22
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Metabolic Associated Fatty Liver Disease; Pancreatic Steatosis; Obese; Lean; Chronic Hepatitis B
MeSH Terms: conditions — Obesity; Hepatitis B, Chronic | interventions — Waist Circumference; Body Mass Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: Obese chronic hepatitis B patients.
  Interventions: Device: Abdominal Ultrasound; Device: Transient elastography; Diagnostic Test: Waist Circumference; Diagnostic Test: Body mass index
- Group II: Lean chronic hepatitis B patients.
  Interventions: Device: Abdominal Ultrasound; Device: Transient elastography; Diagnostic Test: Waist Circumference; Diagnostic Test: Body mass index

INTERVENTIONS:
Device: Abdominal Ultrasound — Standard abdominal ultrasonography performed to evaluate pancreatic steatosis by comparing pancreatic echogenicity to liver and kidney tissue.
Device: Transient elastography — Non-invasive transient elastography used to assess hepatic steatosis and liver stiffness in patients with chronic hepatitis B.
Diagnostic Test: Waist Circumference — The midpoint between the superior aspect of the iliac crests and the lower lateral margins of the ribs using an inelastic tape (TBW Import Ltd) that was 0.5 cm in width and 200 cm in length, according to World Health Organization (WHO) recommendations. Abdominal obesity, determined as a waist circumference of ≥94 cm in males or ≥80 cm in females according to the recommendations of the International Diabetes Federation group
Diagnostic Test: Body mass index — It was calculated by the equation dividing the weight in kilograms by height in meters squared.
  BMI=〖mass〗_kg/(〖height〗_m^2 )

SUMMARY:
This study aimed to evaluate the prevalence of metabolic associated fatty liver disease (MAFLD), fatty pancreas and hepatic fibrosis in obese and lean patients with chronic hepatitis B; either treatment naive or on treatment with first-line nucleos(t)ide analogs.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) infection is one of the major etiologies of chronic liver disease. Pathologies caused by HBV infection range from chronic hepatitis, fibrosis, cirrhosis, to hepatocellular carcinoma (HCC).

Obesity is another significant health burden. Abdominal obesity is a type of obesity that is commonly associated with severe metabolic disorders and cardiovascular diseases.

Previous research has linked abdominal obesity to non-alcoholic fatty liver disease (NAFLD), insulin resistance, type 2 diabetes mellitus (T2DM), and even metabolic syndrome. In 2020, NAFLD was renamed metabolic-associated fatty liver disease (MAFLD) by a group of experts. MAFLD is defined by the presence of liver steatosis in addition to overweight/obesity, type 2 diabetes mellitus (T2DM), or metabolic dysregulation with at least two risk factors, such as an increased waist circumference, pre-diabetes, hypertension, hypertriglyceridemia, and low serum high-density lipoprotein (HDL)-cholesterol levels.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Both sexes.
* Chronic hepatitis B patients.

Exclusion Criteria:

* Hepatitis C virus (HCV) antibody positive.
* Hepatocellular carcinoma (HCC).
* Human immunodeficiency viruses (HIV).
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was carried out in the Tropical Medicine and Infectious Diseases Department, Tanta University.
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Frequency of hepatic steatosis | Immediately post-procedure (Up to 1 hour)
  Frequency of hepatic steatosis (HS) were determined via transient elastography.

SECONDARY OUTCOMES:
Presence of pancreatic steatosis | Immediately post-procedure (Up to 1 hour)
  Presence of pancreatic steatosis was evaluated via ultrasonography.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.